CLINICAL TRIAL: NCT01823055
Title: Safety and Efficacy of a Transvaginal Suture Capturing Mesh Device: The Nordic Uphold LITE Trial
Brief Title: Safety and Efficacy of a Transvaginal Suture Capturing Mesh Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Stockholm County Council, Karolinska Institutet research foundations, Swedish Society of Medicine, Boston Scientific (Unknown)
Responsible Party: Principal Investigator, Daniel Altman, Md, PhD, Associate professor, Karolinska Institutet
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Karolinska Institutet
Record Dates: First submitted 2013-03-28; First posted 2013-04-04 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-03

CONDITIONS: Surgical Repair of Middle Compartment Prolapse (Vaginal Vault or Uterine Prolapse) With or Without Cystocele
MeSH Terms: conditions — Uterine Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Surgery (Experimental): Transvaginal suture capturing mesh device
  Interventions: Procedure: Transvaginal suture capturing mesh device

INTERVENTIONS:
Procedure: Transvaginal suture capturing mesh device — The Uphold™ LITE vaginal support system is an intra-vaginal approach to apical and anterior vaginal wall prolapse repair that utilizes a suture capturing device to place the mesh. After primary dissection the suturing device is used to pull the mesh through the sacrospinous ligament, medial to the ischial spine. An anterior colporraphy was allowed following the Uphold™ LITE procedure at the discretion of the surgeon if deemed necessary.
  Other Names: Uphold™ LITE

SUMMARY:
To perform a clinical safety and efficacy assessment of the Uphold LITE system for pelvic organ prolapse in a prospective multicenter, single cohort study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older and present with primary or recurrent prolapse of the middle vaginal compartment corresponding to stage 2 or higher (according to the Pelvic Organ Prolapse Quantification [POP-Q] system)9,
* with or without anterior vaginal wall prolapse, and
* experiences symptoms of vaginal bulging with or without a previous hysterectomy
* being able to provide oral and written informed consent before entering the study.

Exclusion Criteria:

* previous cancer of any pelvic organ,
* systemic glucocorticoid treatment,
* insulin-treated diabetes,
* an inability to participate in study follow-up or to provide informed consent, or
* the need for any concomitant pelvic surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Immediate and delayed complications related to the surgical procedure | 1 year
  Serious surgical complications are categorised as any surgical event which is potentially life-threatening, internal organ perforation (or other injury), bleeding in excess of 1000 mL or adverse events, related to the surgical procedure, during follow-up which requires re-hospitalisation.

SECONDARY OUTCOMES:
Pelvic Organ Prolapse Quantification system | 1 year
  The secondary efficacy outcome is a composite of objective and subjective measures including POP-Q stage 0 or 1 of the upper vaginal segment (i.e., point C/D, which represents the most distal point of the vaginal apex in relation to the total vaginal length) and a negative response to the question, "Do you experience a feeling of bulging or protrusion in the vaginal area?" (question 16 on the UDI). The secondary outcome measures further include the individual components of the composite end point, other POP-Q measurements and patient-reported urogenital distress.